CLINICAL TRIAL: NCT04660071
Title: Ultrasound Imaging of Quadriceps Muscle in Patients With Knee Osteoarthritis: Reliability of Echo Intensity Measurement
Brief Title: Ultrasound Imaging of Quadriceps Muscle in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERVE KARAPINAR, Research Assisstant, Physiotherapist, Suleyman Demirel University
Other Study IDs: 271
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Reliability,Echo intensity,Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasonographic Assessment, — Ultrasound assessment was performed on rectus femoris (RF), vastus intermedius (VI), vastus medialis (VM) and vastus lateralis (VL) muscles using with an ultrasound-imaging device (Philips Medical Systems EPIQ 5 Release 5.0.2, Amsterdam).
Other: Echo intensity Measurements — All images were analysed using the Image J software (Version 1.48v, National Institutes of Health, Bethesda, MD, USA) by two different analysers (five years and one-year of experience in US image analysis).

SUMMARY:
Echo intensity (EI) assessment using ultrasonography helps monitoring disease-induced muscle quality changes. However, there are no study investigating the reliability of EI in patients with knee osteoarthritis (OA). The primary aim of the present study was to investigate the inter and intra-rater reliability of EI evaluation by grayscale histogram analysis of quadriceps femoris muscle in patients with knee OA. The second aim was to compare the mean grayscale values obtained using both the Free Hand Tool (FHT) and Rectangular Marquee Tool (RMT) methods in ImageJ. Thirty patients with knee OA were included in this cross-sectional study. The echogenicity measurements of the Rectus Femoris, Vastus Inter-medius, Vastus Lateralis and Vastus Medialis were performed by two different researchers. Reliability analysis of EI measurements were calculated with using intraclass correlation coefficient (ICC), standard error of measurement (SEM) and coefficient of variation (CV) and Bland and Altman plot analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients had tibiofemoral joint OA in at least one knee according to the American College of Rheumatology classification criteria with knee pain most days of the past month and osteophytes apparent on knee radiograph were included to the study

Exclusion Criteria:

* Patients were excluded if they had a history of lower limb joint replacement and fracture, rheumatoid arthritis, diabetic neuropathy or polyneuropathy, and cardiovascular and neuromuscular problems.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had tibiofemoral joint OA in at least one knee according to the American College of Rheumatology classification criteria with knee pain most days of the past month, and osteophytes apparent on knee radiograph were included to the study. Patients were excluded if they had a history of lower limb joint replacement and fracture, rheumatoid arthritis, diabetic neuropathy or polyneuropathy, and cardiovascular and neuromuscular problems.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Muscle Echogenicity Assessment ( Physiological parameter) | Thirty minute
  Muscle echogenicity assessed by using ultrasound. Ultrasound assessment was performed on rectus femoris (RF), vastus intermedius (VI), vastus medialis (VM) and vastus lateralis (VL) muscles using with an ultrasound-imaging device (Philips Medical Systems EPIQ 5 Release 5.0.2, Amsterdam). Ultrasound Brightness mode (B-mode) with musculoskeletal scanning and a multi-frequency linear transducer (8-12 MHz, code: eL18-4) were used. For calculating echogenicity of muscles; all images obtained ultrasonography were analysed using the Image J software (Version 1.48v, National Institutes of Health, Bethesda, MD, USA) by two different analysers (five years and one-year of experience in US image analysis). The echogenicity results of the muscles performed by the two researchers recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Karapinar, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No